CLINICAL TRIAL: NCT00004436
Title: Randomized Study of Hormonal Regulation of Infantile Hemangioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Boston Children's Hospital (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13399; CH-B-FDR000967
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-08

CONDITIONS: Hemangioma
Keywords: cardiovascular and respiratory diseases; hemangioma; rare disease
MeSH Terms: conditions — Hemangioma; Respiratory Tract Diseases; Rare Diseases | interventions — Leuprolide; Prednisone

INTERVENTIONS:
Drug: leuprolide
Drug: prednisone

SUMMARY:
OBJECTIVES: I. Evaluate the clinical efficacy of leuprolide, a gonadotropin-releasing hormone agonist (GnRHa), in treating infants with vision-endangering or large, disfiguring hemangiomas.

II. Assess the impact of GnRHa on growth and development during infancy. III. Assess the safety of GnHRa in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo-controlled study. Patients are stratified according to gender and by position of the lesion (periorbital vs nonperiorbital).

All patients receive oral prednisone daily for 3 weeks. Patients are then randomized to receive either placebo or leuprolide IM every 3 weeks, while continuing oral prednisone. Tumors are assessed at 1, 3, and 6 weeks. If the tumor is not responding, the leuprolide will be administered every 2 weeks. Tumors are reassessed at 3 and 6 months, at which point the treatment is stopped. Responding patients are observed every 3 weeks for 3 months. If the tumor begins to grow again, leuprolide may be administered for another 3 months. Patients whose tumors grow rapidly during treatment may crossover to the alternate therapy, repeat the leuprolide or prednisone therapy, or undergo surgical excision.

ELIGIBILITY:
* Presence of hemangioma meeting at least one of the following criteria: Vision-threatening because of induced astigmatism or occlusion of the visual axis or proptosis Severe anatomic distortion compromising function of an organ or creating an unacceptable cosmetic outcome Other complications, e.g., Kasabach-Merritt consumptive coagulopathy, high-output heart failure, etc.
* No lesions that are clearly regressing before therapy
* No vascular malformations other than juvenile hemangiomas

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 1993-07; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Lois Hodgson Smith, Study Chair — Boston Children's Hospital